CLINICAL TRIAL: NCT00943683
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Comparing Montelukast With Placebo in Pediatric Patients Aged 6 to 24 Months With Asthma
Brief Title: Montelukast in Pediatric Patients Aged 6 to 24 Months With Asthma--Safety Study (0476-176)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-176; MK0476-176; 2009_618
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Montelukast
  Interventions: Drug: montelukast sodium
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 4-mg oral granules mixed with applesauce once daily at bedtime for 6 weeks
  Arms: 1
Drug: Comparator: Placebo — Placebo oral granules mixed with applesauce once daily at bedtime for 6 weeks
  Arms: 2

SUMMARY:
A study of Montelukast compared to placebo in asthmatic children aged 6-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in good, stable health
* Patient has been fed solid foods for at least 1 month
* Patients had at least 3 episodes of asthma or asthma-like symptoms, all occurring after 8 weeks of age; at least one within 6 months of the Prestudy Visit
* Patients had to be in need of a controller therapy according to criteria established in the Global Initiative for Asthma (GINA) guidelines

Exclusion Criteria:

* Patient was hospitalized at the start of the study or required a visit to the emergency room due to asthma with in past 2 weeks

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2000-08; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] van Adelsberg J, Moy J, Wei LX, Tozzi CA, Knorr B, Reiss TF. Safety, tolerability, and exploratory efficacy of montelukast in 6- to 24-month-old patients with asthma. Curr Med Res Opin. 2005 Jun;21(6):971-9. doi: 10.1185/030079905X48456. PMID 15969897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 65 study centers in Africa, Asia, Europe, North America, and South America Therapy period: Aug 2000 to Feb 2001
Pre-assignment Details: Patients had at least 3 episodes of asthma or asthma-like symptoms, all occurring after 8 weeks of age; at least one within 6 months of the Prestudy Visit. Patients had to be in need of a controller therapy according to criteria established in the Global Initiative for Asthma (GINA) guidelines
Groups:
- Placebo: Montelukast matching placebo oral granules mixed with applesauce once daily at bedtime for 6 weeks
- Montelukast: Montelukast 4-mg oral granules mixed with applesauce once daily at bedtime for 6 weeks
Period: Overall Study
Arm/Group | Placebo | Montelukast
Started | 81 | 175
Completed | 74 | 169
Not Completed | 7 | 6
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Patient Moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Total
Number analyzed (Participants) | 81 | 175 | 256
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.05 (5.22) | 14.90 (4.70) | 14.63 (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 59 | 81
  Male | 59 | 116 | 175

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinical Adverse Experiences (CAEs) Reported by Patients During the 6-weeks of Treatment
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR'S product, whether or not considered related to the use of the product
Time Frame: During the 6 weeks of treatment
Population: All patients who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 81 | 175
Participants
  With CAEs | 62 | 132
  Without CAEs | 19 | 43

ADVERSE EVENTS:
Time Frame: During the 6 weeks of treatment and including 14 days following treatment
Arm/Group | Placebo | Montelukast
Serious Adverse Events (participants affected / at risk) | 1/81 | 7/175
Other Adverse Events (participants affected / at risk) | 55/81 | 112/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Montelukast (N=175)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Drug Overdose (Injury, poisoning and procedural complications) | 0 | 1
Inguinal Hernia (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Aspiration (Condition) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Montelukast (N=175)
Fever (General disorders) | 11 | 23
Upper Respiratory Infection (Infections and infestations) | 17 | 56
Diarrhea (Gastrointestinal disorders) | 10 | 18
Vomiting (Gastrointestinal disorders) | 9 | 15
Conjunctivitis (Eye disorders) | 5 | 4
Otitis Media (Ear and labyrinth disorders) | 5 | 15
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 | 14
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 | 32
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.